CLINICAL TRIAL: NCT02161510
Title: A Multiple Dose Study to Evaluate Safety, Pharmacokinetics, and Pharmacodynamics of MK-2248 in Subjects With Hepatitis C Infection
Brief Title: Safety, Pharmacokinetics, and Pharmacodynamics of MK-2248 in Participants With Hepatitis C (MK-2248-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2248-002; 2014-001494-14 (EudraCT Number)
Record Dates: First submitted 2014-06-10; First posted 2014-06-11 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- Part I: MK-2248 200 mg (Panel A) (Experimental): HCV participants will take MK-2248 200 mg by mouth once daily for 7 days.
  Interventions: Drug: MK-2248
- Part I: MK-2248 ≤800 mg (Panel B) (Experimental): Based on safety, PK, and PD data from the preceding panel, HCV participants will take MK-2248 at approximately ≤800 mg by mouth once daily for 7 days.
  Interventions: Drug: MK-2248
- Part I: MK-2248 ≤800 mg (Panel C) (Experimental): Based on safety, PK, and PD data from the preceding panel, HCV participants will take MK-2248 at approximately ≤800 mg by mouth for 7 days.
  Interventions: Drug: MK-2248
- Part I: MK-2248 ≤800 mg (Panel D) (Experimental): Based on safety, PK, and PD data from the preceding panel, HCV participants will take MK-2248 at approximately ≤800 mg by mouth once daily for 7 days.
  Interventions: Drug: MK-2248
- Part II: MK-2248 200 mg (Panel E) (Experimental): HCV participants will take MK-2248 200 mg by mouth once daily for 7 days.
  Interventions: Drug: MK-2248
- Part II: MK-2248 ≤800 mg (Panel F) (Experimental): Based on safety, PK, and PD data from the preceding panel, HCV participants will take MK-2248 at approximately ≤800 mg by mouth once daily for 7 days.
  Interventions: Drug: MK-2248
- Part II: MK-2248 ≤800 mg (Panel G) (Experimental): Based on safety, PK, and PD data from the preceding panel, HCV participants will take MK-2248 at approximately ≤800 mg by mouth once daily for 7 days.
  Interventions: Drug: MK-2248
- Part II: MK-2248 ≤800 mg (Panel H) (Experimental): Based on safety, PK, and PD data from the preceding panel, HCV participants will take MK-2248 at approximately ≤800 mg by mouth once daily for 7 days.
  Interventions: Drug: MK-2248
- Part III: MK-2248 ≤800 mg (Panel I) (Experimental): Based on safety, PK, and PD data from the preceding panel, HCV participants will take MK-2248 at approximately ≤800 mg by mouth once daily for 7 days.
  Interventions: Drug: MK-2248
- Part III: MK-2248 ≤800 mg (Panel J) (Experimental): Based on safety, PK, and PD data from the preceding panel, HCV participants will take MK-2248 at approximately ≤800 mg by mouth once daily for 7 days.
  Interventions: Drug: MK-2248

INTERVENTIONS:
Drug: MK-2248 — MK-2248 in once-daily oral doses of 200-≤800 mg for 7 days

SUMMARY:
The objective of this study is to identify a safe dose of MK-2248 in participants with Hepatitis C Virus (HCV) that mediates at least a 3 log10 reduction in viral load (VL) from baseline. It is anticipated that once-daily administration of a safe and well tolerated dose of MK-2248 will reduce VL by at least 3 log10 IU/mL.

DETAILED DESCRIPTION:
In this Phase 1b study, the pharmacokinetic (PK), pharmacodynamic (PD), and safety profile of MK-2248 in HCV-infected participants will be evaluated as follows: Part I will assess sequentially ascending MK-2248 doses from 200 mg to ≤800 mg over 4 panels (A, B, C, and D). Part II will assess sequentially ascending MK-2248 doses from 200 mg to ≤800 mg over 4 panels (E, F, G, and H). Part III will assess sequentially ascending MK-2248 doses ranging up to ≤800 mg in 2 panels (I and J). The potential relationship between plasma MK-2248 levels and VL reduction will be determined.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of chronic HCV defined by positive serology for HCV or positive HCV RNA for at least 6 months and detectable HCV RNA in peripheral blood ≥10^5 IU/mL at screening
* Body Mass Index (BMI) ≥18 to <37 kg/m^2
* in good health other than HCV infection with normal laboratory values

Exclusion Criteria:

* history of clinically significant and not stably controlled endocrine, gastrointestinal, cardiovascular, hematological, hepatic (excepting HCV infection), immunological, renal, respiratory, genitourinary, or major neurological abnormalities or disease
* history of cancer other than adequately treated non-melanomatous skin carcinoma, malignancies which have been successfully treated ≥10 years prior with no recurrence, or cancer that is unlikely to sustain a recurrence for the duration of the trial
* history of significant multiple and/or severe allergies or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* positive for hepatitis B surface antigen or human immunodeficiency virus
* had major surgery or lost 1 unit of blood within 4 weeks prior to screening
* QTc interval ≥470 msec (males) or ≥480 msec (females)
* received prior treatment with other HCV inhibitors
* clinical or laboratory evidence of decompensated liver disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-07; Primary Completion 2014-11 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Maximum change from baseline in VL | Up to Day 42
Number of participants experiencing an adverse event (AE) | Up to Day 42
Number of participants who discontinue from study treatment due to an AE | Up to Day 7

SECONDARY OUTCOMES:
Plasma concentration at 24 hours post-dose (C24hr) of MK-2248 and circulating metabolite(s) | Up to Day 10
Area under the plasma-concentration curve at zero to 24 hours post-dose (AUC[0-24hr]) of MK-2248 and circulating metabolite(s) | Up to Day 10
Maximum observed post-dose plasma concentration (Cmax) of MK-2248 and circulating metabolite(s) | Up to Day 10
Time post-dose at which the maximum observed plasma concentraton (Tmax) of MK-2248 and circulating metabolite(s) occurs | Up to Day 10
Time required for Cmax to decrease by half (apparent t1/2) of MK-2248 and circulating metabolite(s) in plasma | Up to Day 10
Accumulation ratio of MK-2248 and circulating metabolite(s) in plasma | Up to Day 10
Total clearance (amount of drug cleared relative to the total systemically available amount per unit time [CL/F]) of MK-2248 in plasma | Up to Day 10
Apparent volume of distribution (V/F) of MK-2248 in plasma | Up to Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC